CLINICAL TRIAL: NCT04187976
Title: Peripheral Eosinophils Phenotypes in Airway Inflammatory Diseases: Towards Proper Clustering and Therapeutic Targeting
Brief Title: Eosinophils Endotypes in Chronic Airway Inflammatory Diseases
Acronym: PLEIAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_81; 2019-A01457-50 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Eosinophilic Asthma; Chronic Sinusitis; Eosinophilic Rhinitis
Keywords: Eosinophil; asthma; chronic rhinosinusitis with nasal polyps; biotherapy; endotype
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Eosinophils from blood samples,nasal polyps and induced sputum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with moderate to severe uncontrolled asthma: Patients with moderate to severe uncontrolled asthma defined on clinical assessment and spirometric criteria. Non controlled asthma is considered when ACQ score ≥ 1.5 or in case of acute exacerbation
- Patients with recalcitrant CRSwNP requiring sinus surgery: The medical failure in CRSwNP is defined as persistent disease in spite of 3 courses of oral corticosteroid and double dose of local corticoid over 12 months
- Patients with concomitant CRSwNP and uncontrolled asthma: Patients with concomitant CRSwNP and moderate to severe uncontrolled asthma
- Healthy subjects: Patients without any airway inflammatory disease or atopy

SUMMARY:
Asthma and chronic rhinosinusitis with nasal polyps (CRSwNP) are frequently described as unified airway inflammatory diseases. Both heavily impacts quality of life with substantial productivity loss. They share the same pathophysiologic pattern based upon proTh2 immune response with blood eosinophils recruitment. Eosinophils are the major actor of persistent mucosal inflammation by promoting their own survival, by attracting other inflammatory cells and by producing cytotoxic proteins involved in mucosal remodeling.

Promising anti-Th2 therapeutic approaches (i.e.anti-IgE, anti-interleukin 5 (IL-5), anti-IL-4, anti-IL-13) are considered as effective alternative options to long-term corticosteroid treatment. Their advantage in recalcitrant CRSwNP is under consideration. Moreover, we still need to delineate the good responders to improve theirs indications.

The objective is to assess blood eosinophil immunophenotypes in asthma or CRSwNP. Flow cytometric expression of activation markers on eosinophil membrane will be compared with a group of healthy subjects. Innovative data on eosinophil involvement in airway diseases will be obtained. The major outcome will be to depict patients' endotypes for a better selection of immunotherapies.

ELIGIBILITY:
Inclusion Criteria:

For all groups:

* Social insured patient
* Patient willing to comply with all procedures of the study and its duration
* Provision of signed and dated informed consent form prior to any study specific procedure

For Group 1:

- Patients with moderate to severe uncontrolled asthma, confirmed by relevant clinical symptoms and proven variable airway obstruction, and assessed by an expert pulmonologist according to spirometry criteria (absolute and weighed Forced Expiratory Volume (FEV) and Forced Vital Capacity (FVC) before and after 2 test),(see CRF for details). Uncontrolled asthma will be defined by an ACQ score ≥ 1.5. or acute exacerbation

For Groups 2 and 3:

* Patients with medically refractory bilateral sino-nasal polyposis requiring sinus surgery, according to an expert rhinologist. CRSwNP diagnosis is based on the presence of bilateral nasal polyps from both side of middle turbinates on nasoendoscopy and bilateral sinus opacification on CT scan. Briefly, CRSwNP is considered as refractory when symptoms are still not controlled after 3 courses of oral corticosteroid and double dose of nasal corticosteroid during the last 12 months
* Patients with both uncontrolled asthma and recalcitrant CRSwNP with or without concomitant aspirin-exacerbated respiratory disease (AERD) (group 3)

For Group 4:

- Healthy subjects without any airway disease or any atopic status, as assessed by a questionnaire and a medical examination

Exclusion Criteria:

For all groups:

* Patients with any other form of secondary CRSwNP (eg, cystic fibrosis, primary ciliary dyskinesia).
* Patients with any form of secondary severe asthma (eg (non)eosinophilic granulomatosis with polyangiitis, allergic bronchopulmonary aspergillosis)
* Patients taking or having taken systemic corticosteroid, leukotriene receptor antagonist, theophylline or long-term macrolide therapy within 1 month prior to sample collections, anti-immunoglobulin E therapy (omalizumab) anti-IL-5/5R or anti IL-4R/anti-IL13 therapies within 6 months before inclusion
* Patients followed up for another inflammatory or auto-immune disease
* Previous allogeneic bone marrow transplant
* Patients with ongoing sub-cutaneous or sub-lingual anti-allergenic immunotherapies
* Patients with active smoking or history of smoking > 10 packages-year for asthma patients
* Pregnant, breastfeeding, or lactating women
* Non-coverage by the social security insurance
* Patient unable to receive informed information
* Refusal to sign the consent form
* Unwillingness or inability to follow the study procedures, in the opinion of the investigator
* Person deprived of the liberty
* Person benefiting from a system of legal protection (guardianship…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients for the study will be targeted either during hospitalization in Pneumology for uncontrolled asthma patients, during ENT visit for scheduling of sinus surgery (recalcitrant CRSwNP).
  The healthy subjects are going to be screened in the Clinical Investigation Center of the University Hospital of Lille. Subjects will be contacted by phone after selection in the database.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of blood eosinophils with expression of CD69 marker in patients with uncontrolled asthma alone, recalcitrant chronic rhinosinusitis with nasal polyps (CRSwNP) alone, uncontrolled asthma and recalcitrant CRSwNP and in healthy subjects. | Baseline
  CD69 expression is measured with flow cytometry on blood eosinophils cell surface.
  The percentage of blood eosinophils positive for CD69 is compared between the four groups of patients (uncontrolled asthma alone, recalcitrant CRSwNP alone, uncontrolled asthma and recalcitrant CRSwNP and in healthy subjects)

SECONDARY OUTCOMES:
Percentage of blood eosinophils with expression of HLADR marker in patients with uncontrolled asthma alone, recalcitrant CRSwNP alone, uncontrolled asthma and recalcitrant CRSwNP and in healthy subjects. | baseline
  HLADR expression is measured with flow cytometry on blood eosinophils cell surface.
  The percentage of blood eosinophils positive for HLADR is compared between the four groups of patients (uncontrolled asthma alone, recalcitrant CRSwNP alone, uncontrolled asthma and recalcitrant CRSwNP and in healthy subjects)
Percentage of activated blood eosinophils in patients with uncontrolled asthma alone, recalcitrant CRSwNP alone, uncontrolled asthma and recalcitrant CRSwNP and in healthy subjects. | baseline
  Activated status of blood eosinophils is based on concomittant expression of biomarkers ( CD69, HLADR, CCR3) with flow cytometry. The percentage of activated blood eosinophils is compared between the four groups of patients (uncontrolled asthma alone, recalcitrant CRSwNP alone, uncontrolled asthma and recalcitrant CRSwNP and in healthy subjects).
Comparison of the percentage of activated eosinophils in blood with the percentage of activated eosinophils in induced sputum in uncontrolled asthma (with or without CRSwNP). | baseline
  Activated status of eosinophils in blood and in induced sputum is based on concomittant expression of biomarkers ( CD69, HLADR, CCR3) with flow cytometry.
Comparison of the percentage of activated eosinophils in blood with the percentage of activated eosinophils in nasal polyps in CRSwNP patients (with or without uncontrolled asthma). | baseline
  Activated status of eosinophils in blood and in nasal polyps is based on concomittant expression of biomarkers ( CD69, HLADR, CCR3) with flow cytometry.
Comparison of qualitative transcriptomic profiles of blood eosinophils in patients with uncontrolled asthma alone, recalcitrant chronic rhinosinusitis with nasal polyps (CRSwNP) alone, uncontrolled asthma and recalcitrant CRSwNP. | baseline
  Transcriptomic profiles will be compared between CRSwNP with or without uncontrolled asthma and between uncontrolled asthma with or without CRSwNP.
  A two-fold differential expression will be used for comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Chenivess, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU Lille, Lille, France